CLINICAL TRIAL: NCT01154959
Title: Characterization of Immune Responses in Treatment-induced Latency in Pulmonary Tuberculosis
Brief Title: Latency in Pulmonary Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dr. S. Subash Babu, Scientific Director, NIH-NIRT-ICER, Tuberculosis Research Centre, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTB01
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Tuberculosis
Keywords: Pulmonary TB; Immune response; ATT; Immune responses in pulmonary tuberculosis; Predictors for relapse
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Moxifloxacin; Isoniazid; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Regimen 1 (Experimental): Rifampicin, isoniazid, pyrazinamide, ethambutol and moxifloxacin daily for 3 months (3RHZEM)
  Interventions: Drug: Moxifloxacin, Isoniazid, Rifampicin Pyrazinamide, Ethambutol
- Regimen 2 (Experimental): Rifampicin, isoniazid, pyrazinamide, ethambutol and moxifloxacin daily for 2 months followed by rifampicin, isoniazid, and moxifloxacin daily for 2 months (2 RHZEM daily / 2 RHM daily)
  Interventions: Drug: Moxifloxacin, Isoniazid, Rifampicin Pyrazinamide, Ethambutol
- Regimen 3 (Experimental): Rifampicin, isoniazid, pyrazinamide, ethambutol and moxifloxacin daily for 2 months followed by rifampicin, isoniazid, and moxifloxacin thrice weekly for 2 months (2 RHZEM daily / 2RHM thrice weekly)
  Interventions: Drug: Moxifloxacin, Isoniazid, Rifampicin Pyrazinamide, Ethambutol
- Regimen 4 (Experimental): Rifampicin, isoniazid, pyrazinamide, ethambutol and moxifloxacin daily for 2 months followed by rifampicin, isoniazid, ethambutol and moxifloxacin thrice weekly for 2 months (2 RHZEM daily / 2 RHEM thrice weekly)
  Interventions: Drug: Moxifloxacin, Isoniazid, Rifampicin Pyrazinamide, Ethambutol
- Control Regimen (Active Comparator): Rifampicin, isoniazid, pyrazinamide and ethambutol thrice weekly for 2 months followed by rifampicin and isoniazid thrice weekly for 4 months (2 RHZE thrice weekly / 4 RH thrice weekly)
  Interventions: Drug: Moxifloxacin, Isoniazid, Rifampicin Pyrazinamide, Ethambutol

INTERVENTIONS:
Drug: Moxifloxacin, Isoniazid, Rifampicin Pyrazinamide, Ethambutol — Moxifloxacin (400mg), Isoniazid (300mg daily, 600mg thrice weekly), Rifampicin (450mg, and 600mg for patients weighing 60kg or more), Pyrazinamide (1500mg), Ethambutol (800mg)

SUMMARY:
The immune responses in latent tuberculosis are poorly understood. While it is difficult to define the onset of latency during natural infection, patients undergoing treatment for tuberculosis are driven into a state of latency or cure. The present study on the effect of 3 and 4 month regimens containing moxifloxacin in sputum smear and culture positive pulmonary tuberculosis (TRC Study number 24) offers us the opportunity to study definitive immune responses pre and post treatment. We will evaluate a variety of innate and adaptive immune responses in patients before and after treatment and our study will compare the differences in immuno-phenotype (eg. Markers of T, B and NK cell activation, proliferation and regulatory phenotype) and function (eg. Production of cytokines, proliferative responses to TB antigens) at different time points following treatment. In addition, since a small percentage of patients will undergo relapse following treatment, the kinetics of immune responses in these patients will used to assess immunological predictors of relapse in tuberculosis.

DETAILED DESCRIPTION:
Although Mycobacterium tuberculosis (Mtb) infects approximately 2 billion people worldwide, 90% of Mtb infected individuals are able to resist overt disease (active tuberculosis) development and manifest only latent infection. Latent tuberculosis (TB) is defined as the persistent presence of live Mtb within an infected host without causing disease. It is characterized by a delayed type hypersensitivity response to purified protein derivative (PPD) mediated by mycobacteria specific T cells. During latency, Mtb is contained in localized granulomas where the mycobacteria reside in macrophages and in which growth and replication appears to be constrained. Maintenance of the granulomatous lesion is mediated by CD4+ and CD8+ T cells. Based on murine models, immunity to Mtb requires Th1 responses and (to a lesser extent) Th17 responses. Thus, IL 12, IFN gamma, and TNF alpha (and IL 17 and IL 23) all play important roles in induction and maintenance of protective immune responses against tuberculous disease. Although CD4+ T lymphocytes of Th1 type are critical for protective immunity, evidence exists that CD8+ T cells as well as unconventional T cells (gamma-delta T cells and CD 1 restricted T cells) contribute to optimum protection in susceptible animal models. Aside from producing cytokines that activate macrophages and initiate granuloma formation, T cells also have direct mycobactericidal activities through the concerted actions of perforins and granulysins.

T cell differentiation into Th1 and Th2 lineages based on their cytokine profile and transcription factor expression has served as the basis of our understanding the pathogenesis of a variety of infectious and allergic diseases. With the advent of newer techniques, T cell differentiation has expanded into several subsets, including Tregs, Th17 cells, and polyfunctional T cells, among others. Th1 cells are absolutely essential for resistance to TB both in mice and humans. Deficiencies in the IL 12 IFN gamma Stat1 pathway leads to disseminated mycobacterial infection in humans and to abrogation of resistance in mice. In addition, TNF alpha, another Th1 cytokine, is of almost equal importance, as treatment with biologics (e.g., anti TNF alpha antibodies) for inflammatory disorders such as rheumatoid arthritis has caused reactivation of TB in some individuals.

Latent TB can be maintained for the lifetime of the individual unless the immunological balance between the host and the pathogen is perturbed, resulting in reactivation of Mtb and active disease. The host and environmental factors involved in compromising the ability to contain latent infection are human immunodeficiency virus co infection, malnutrition, aging, stress, Type 2 diabetes, use of immunosuppressive agents, and other genetic factors. On the pathogen side, latency is thought to reflect a transition from replicating to nonreplicating dormant bacilli, with this transition being influenced by a variety of factors including oxygen deprivation and nitric oxide. The use of in vitro and in vivo models of latency combined with genome wide transcriptome profiling has led to the identification of Mtb genes highly expressed during latency called dosR or devR (dormancy) genes; however, each of the host and pathogen related factors controlling resistance and/or susceptibility to TB awaits complete elucidation.

The subsets of CD4+ T cells constitute an ever expanding repertoire, classified by their discrete cytokine profiles and often by expression of prototypical transcription factors and/or cell surface molecules. Two relatively newly emerging CD4+ T cell subsets of importance are Th17 cells, characterized by production of IL 17 family of cytokines, and regulatory T cells (Tregs), characterized by surface expression of CD25 and the transcription factor FoxP3. Little is known about the role of these two subsets in latent TB. The mechanism by which Mtb subverts immune responses to establish chronic, latent infection is also not well understood. Recently, a number of regulatory factors, including Tregs, IL 10, TGF-beta, CTLA 4, and PD 1, have been implicated in the establishment of chronic viral, bacterial, and parasitic infections.

The role of T, B and NK cells in the evolution of the immune response following therapy in Mycobacterium tuberculosis infection has to be elucidated. The development of cellular immune responses in TB-infected patients post-chemotherapy to delineate the cellular arms of immunity in response to crude and defined TB antigens in treated patients needs to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Residing in or around Chennai or Madurai
* No anti-TB treatment in the past or should have had less than one month of treatment (but less than one week in the preceding one month before enrollment in the study)
* At least two sputum smears should be positive for tubercle bacilli by fluorescent microscopy
* Express willingness to attend the treatment centre for supervised treatment
* Express willingness for home visits by the staff of the centre
* Express willingness to give written informed consent

Exclusion Criteria:

* Body weight less than 30 kg
* Hepatic or renal disease as evidenced by clinical or biochemical abnormalities
* Diabetes mellitus
* A history of seizure or loss of consciousness
* Psychiatric illness
* An abnormal electrocardiogram or anti-arrhythmic medication
* Those in a moribund state
* Sero-positive for HIV antibodies
* Pregnancy or lactation
* Visual disorders other than refractory error

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The immune response to crude antigens - PPD and CFA and defined antigens - ESAT-6 and CFP-10 as well as positive controls- SEB and anti-CD3. | 2 years

SECONDARY OUTCOMES:
Determining the correlation of increase in regulatory factors with the development of relapse in treated TB patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Subash Babu, MBBS, PhD, Principal Investigator — Tuberculosis Research Centre, India
Locations (1):
- Tuberculosis Research Centre, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Comstock GW, Livesay VT, Woolpert SF. The prognosis of a positive tuberculin reaction in childhood and adolescence. Am J Epidemiol. 1974 Feb;99(2):131-8. doi: 10.1093/oxfordjournals.aje.a121593. No abstract available. PMID 4810628
- [Background] Lillebaek T, Dirksen A, Baess I, Strunge B, Thomsen VO, Andersen AB. Molecular evidence of endogenous reactivation of Mycobacterium tuberculosis after 33 years of latent infection. J Infect Dis. 2002 Feb 1;185(3):401-4. doi: 10.1086/338342. Epub 2002 Jan 17. PMID 11807725
- [Background] Wayne LG, Sohaskey CD. Nonreplicating persistence of mycobacterium tuberculosis. Annu Rev Microbiol. 2001;55:139-63. doi: 10.1146/annurev.micro.55.1.139. PMID 11544352
- [Background] EDWARDS PQ, EDWADS LB. Story of the tuberculin test from an epidemiologic viewpoint. Am Rev Respir Dis. 1960 Jan;81(1)Pt 2:1-47. No abstract available. PMID 13819440
- [Background] Kaufmann SH. How can immunology contribute to the control of tuberculosis? Nat Rev Immunol. 2001 Oct;1(1):20-30. doi: 10.1038/35095558. PMID 11905811
- [Background] Lin MY, Ottenhoff TH. Not to wake a sleeping giant: new insights into host-pathogen interactions identify new targets for vaccination against latent Mycobacterium tuberculosis infection. Biol Chem. 2008 May;389(5):497-511. doi: 10.1515/bc.2008.057. PMID 18953716
- [Background] Ulrichs T, Kaufmann SH. New insights into the function of granulomas in human tuberculosis. J Pathol. 2006 Jan;208(2):261-9. doi: 10.1002/path.1906. PMID 16362982
- [Background] Khader SA, Cooper AM. IL-23 and IL-17 in tuberculosis. Cytokine. 2008 Feb;41(2):79-83. doi: 10.1016/j.cyto.2007.11.022. Epub 2008 Jan 22. PMID 18218322
- [Background] North RJ, Jung YJ. Immunity to tuberculosis. Annu Rev Immunol. 2004;22:599-623. doi: 10.1146/annurev.immunol.22.012703.104635. PMID 15032590
- [Background] Locht C, Rouanet C, Hougardy JM, Mascart F. How a different look at latency can help to develop novel diagnostics and vaccines against tuberculosis. Expert Opin Biol Ther. 2007 Nov;7(11):1665-77. doi: 10.1517/14712598.7.11.1665. PMID 17961090
- [Background] Murphy KM, Reiner SL. The lineage decisions of helper T cells. Nat Rev Immunol. 2002 Dec;2(12):933-44. doi: 10.1038/nri954. PMID 12461566
- [Background] Dong C. TH17 cells in development: an updated view of their molecular identity and genetic programming. Nat Rev Immunol. 2008 May;8(5):337-48. doi: 10.1038/nri2295. PMID 18408735
- [Background] McGeachy MJ, Cua DJ. Th17 cell differentiation: the long and winding road. Immunity. 2008 Apr;28(4):445-53. doi: 10.1016/j.immuni.2008.03.001. PMID 18400187
- [Background] Weaver CT, Hatton RD, Mangan PR, Harrington LE. IL-17 family cytokines and the expanding diversity of effector T cell lineages. Annu Rev Immunol. 2007;25:821-52. doi: 10.1146/annurev.immunol.25.022106.141557. PMID 17201677
- [Background] Fontenot JD, Rudensky AY. Molecular aspects of regulatory T cell development. Semin Immunol. 2004 Apr;16(2):73-80. doi: 10.1016/j.smim.2003.12.002. PMID 15036230
- [Background] Sakaguchi S. Naturally arising CD4+ regulatory t cells for immunologic self-tolerance and negative control of immune responses. Annu Rev Immunol. 2004;22:531-62. doi: 10.1146/annurev.immunol.21.120601.141122. PMID 15032588
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Li MO, Flavell RA. Contextual regulation of inflammation: a duet by transforming growth factor-beta and interleukin-10. Immunity. 2008 Apr;28(4):468-76. doi: 10.1016/j.immuni.2008.03.003. PMID 18400189
- [Derived] Kumar NP, Moideen K, Dhakshinraj SD, Banurekha VV, Nair D, Dolla C, Kumaran P, Babu S. Profiling leucocyte subsets in tuberculosis-diabetes co-morbidity. Immunology. 2015 Oct;146(2):243-50. doi: 10.1111/imm.12496. Epub 2015 Jul 6. PMID 26095067
- [Derived] Kumar NP, Sridhar R, Nair D, Banurekha VV, Nutman TB, Babu S. Type 2 diabetes mellitus is associated with altered CD8(+) T and natural killer cell function in pulmonary tuberculosis. Immunology. 2015 Apr;144(4):677-86. doi: 10.1111/imm.12421. PMID 25363329